CLINICAL TRIAL: NCT07306091
Title: Ultrasound-guided Decannulation With Critically Ill Patients; a Prospective Cohort Study
Brief Title: Decanulation in Critically Ill Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Pınar Küçükdemirci Kaya, associated proffesor, Uludag University
Other Study IDs: BursaUludag ( 2024-10/15)
Record Dates: First submitted 2025-11-17; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Decanulation
Keywords: Ultrasound; decanulation; critically illness; weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suitable for decannulation after tracheostomy within the specified date range: Patients who were deemed suitable for decannulation after tracheostomy within the specified date range and who underwent FEES by an otolaryngologist
  Interventions: Device: ultrasound guided airway examination

INTERVENTIONS:
Device: ultrasound guided airway examination — the position of the vocal cords (right, left, cadaveric, normal), movements with phonation and respiration, and vocal fold displacement velocity (VFDV) to control air permeability will be measured by bedside ultrasound by deflating the cuff of the tracheostomy cannula, the cannula will be removed and the same measurements will be taken again with ultrasonography, before being transferred to the otolaryngology clinic (OT) for Flexible Endoscopic Evaluation of Swallowing (FEES) exam

SUMMARY:
Purpose of the Study: To predict potential problems (such as shortness of breath and obstruction of the airway due to vocal cord immobility) before the tracheostomy cannula is removed, the patient's vocal cords, their movement, and airflow rate will be assessed at the bedside. The patient will also be examined using routine methods to identify these problems, and the results will be compared with ultrasound scans. The study aims to determine the success and failure of ultrasound in detecting these problems. Method and Procedures: While the patient is receiving treatment in the intensive care unit, the probe of the existing ultrasound device will be placed on the patient's neck, over the cannula, and the movement of the vocal cords and airflow rate will be assessed.

DETAILED DESCRIPTION:
In this study, in patients who will be treated in our intensive care unit between 01.07.2024 and 01.12.2025 and who are deemed suitable for decannulation after tracheostomy [patients must be clinically stable, have been able to stay off the ventilator for at least 48 hours and have appropriate arterial blood gases taken during this time, have no dyspnea, GCS>10, have swallowing and cough reflexes, have no problems with mouth opening, and have secretions less than 1/3 of the length of a catheter (1)], the position of the vocal cords (right, left, cadaveric, normal), movements with phonation and respiration, and vocal fold displacement velocity (VFDV) to control air permeability will be measured by bedside ultrasound by deflating the cuff of the tracheostomy cannula, the cannula will be removed and the same measurements will be taken again with ultrasonography, before being transferred to the otolaryngology clinic (OT) for Flexible Endoscopic Evaluation of Swallowing (FEES) exam. The accuracy of the measurement will be confirmed by two researchers by video recording, and the findings will be compared with the FEES examination. Additionally, demographic characteristics, comorbidities, acute physiology and chronic health assessment scores (APACHEII), sequential organ failure assessment score (SOFA), comorbidities, decannulation failure (repeat tracheostomy or intubation within 2 days after decannulation) and prognosis (90 day-mortality) after decanulation will be recorded for patients meeting the above criteria.

ELIGIBILITY:
Inclusion Criterias

1. Critically ill patients (CIPs) who are receiving treatment within the specified time period and who require a tracheostomy.
2. Critically ill patients who are suitable for decannulation (underwent spontaneous breathing trials with the use of CPAP ( CPAP level of maximum 6 cm of water and maximum 10 cm of water pressure support at least 24 hours ).
3. Critically ill patients with intact swallowing reflexes ( patients were first examined for GAG reflexes, followed by ultrasonography; changes in muscle length and contraction velocity during swallowing were measured in a sagittal section using a convex probe ,
4. CIPs with GCS>8.

Exclusion Criteria:

1.Critically ill patients under 18 years of age. 2.Critically ill patients who do not require tracheostomy. 3.Critically ill patients who are spontaneously breathing and can be weaned off the ventilator for <24 hours 4.Critically ill patients with GCS < 8. 5.Critically ill patients with absent swallowing reflexes

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients whom suitable for decanulation after tracheostomy
Sampling Method: Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Airway examination with ultrasound for decanulation | 15 months
  This study aimed to observe at what doppler velocity values (cm/s) successful decannulation (168 hours without ventilation) could be achieved in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag Universty Faculty of MedicineDepartment of Anesthesiology and Reanimation, Bursa, Turkey, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Informed Consent Form (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT07306091/ICF_000.pdf